CLINICAL TRIAL: NCT04413968
Title: Contamination and Transmission of the SARS-CoV-2 Virus in Exposed, Confined and Community-based Infants: A Cross-sectional, Multicentre, Interventional Seroprevalence Study
Brief Title: COVID-19 Infection and Transmission in Exposed, Confined and Community-based Infants
Acronym: COVIDOCRECHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP200587; 2020-A01540-39 (Other: Registry ID : IDRCB)
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-05

CONDITIONS: Coronavirus; Coronavirus Infection; Covid19; Sars-CoV2
Keywords: Nursery; Child
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: Cross-sectional, multi-center, non-randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): nasopharyngeal and blood sample
  Interventions: Diagnostic Test: Rapid detection test; Diagnostic Test: Nasopharyngeal swab; Diagnostic Test: Stool collection

INTERVENTIONS:
Diagnostic Test: Rapid detection test — Rapid serological test by taking 3 drops of blood from the fingertip via the TDR device (rapid detection test) for children, supervising nursery staff and hospital laboratory and administrative staff
Diagnostic Test: Nasopharyngeal swab — Posterior nasopharyngeal swabbing in children
Diagnostic Test: Stool collection — Stool collection in children

SUMMARY:
According to epidemiological models, the seroprevalence of SARS-CoV-2 infection in Île-de-France as of 11 May was between 10 and 15%. Preliminary data on the number of professionals evicted from nurseries on suspicion of COVID-19 (on clinical grounds) seem to be of the same order of magnitude, but need to be confirmed by a biological technique. Children would be susceptible to infection but often asymptomatic.

DETAILED DESCRIPTION:
SARS-CoV-2, an emerging respiratory virus of the coronavirus family, is responsible for a global pandemic of which Europe has become the epicentre. Infection with the virus causes a disease called COVID-19, whose expression most often includes cough, fever, fatigue, myalgia, anosmia, ageusia and gastrointestinal symptoms, and which can be complicated by severe pneumonia requiring resuscitation and which can lead to death. Morbidity and mortality are clearly age-related and while illness and hospitalisations occur in all age groups, deaths occur mostly in the older age groups.

In the absence of curative treatment and vaccination, the only real measures capable of slowing the progression of the disease are large-scale social distancing measures. In analogy to community-based viral epidemics such as seasonal influenza, children were initially considered a potential vector of transmission, which led to the preventive measure of school closures. In France, this closure came into force on 14 March 2020.

Children are considered to be little affected by the coronavirus-19 epidemic because even if screening strategies differ, they represent less than 3% of the cases confirmed in the various studies.

In a period of confinement and reduction in the number of children cared for, in a crèche for children of healthcare workers, in a context of proximity and high risk of cross transmission, the frequency of symptomatic and asymptomatic forms of SARS-Cov-2 in children and staff would be comparable to the general population.

We hypothesize a susceptibility to infection in children but low transmission, which should lead to a cumulative prevalence of infection among daycare staff comparable to that obtained in a sample of professionals who do not come into contact with children in their work (here hospital laboratory and administrative staff).

ELIGIBILITY:
Inclusion Criteria:

Population 1 :

* Children of priority staff welcomed in the crèche during the period of confinement, i.e. from 15 March to 9 May, regardless of the length of time they are in the crèche during this period and their "symptomatic or not" status during this period or on the day of inclusion.
* Consent of the holders of parental authority
* Affiliated to a social security system or entitled person

Population 2 :

* Nursery staff, regardless of their status/occupation and having had contact with the children during the period of confinement regardless of how long they have been in the nursery during this period and their "symptomatic or not" status during this period or on the day of inclusion.
* Consent to participate
* Affiliated to a social security system or entitled person

Population 3 :

* Hospital staff not exposed to patients and/or children, with or without children in day care, working in the bacteriology, biochemistry and biological haematology laboratories or in an administrative department of the participating hospitals.
* Affiliated to a social security system or entitled person

Exclusion Criteria:

Population 1 :

* Refusal to sign consent by parents
* Clinical condition requiring urgent medical assessment (attending physician or transfer to paediatric emergency)

Population 2 and 3 :

* Refusal to sign consent for staff
* Clinical condition requiring urgent medical evaluation

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Assess the serological status/rate of past infections in the children of priority staff in the nursery during the containment period | Day of intervention (1 day)
  Proportion of children with a positive rapid serological test (presence of anti-SARS-CoV2 antibodies (IgM or IgG)).

CONTACTS AND LOCATIONS:
Overall Officials: Eric LACHASSINNE, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (11):
- France (11):
  - Hopital Avicenne, Bobigny
  - Hôpital Jean Verdier - Service de Pédiatrie, Bondy
  - Hôpital Jean Verdier, Bondy
  - Hôpital Antoine béclère, Clamart
  - Hôpital Louis Mourier, Colombes
  - CH intercommunal de Créteil, Créteil
  - Hôpital Annecy Genevois, Épagny
  - Hôpital Andé Mignot, Le Chesnay
  - Hôpital Trousseau, Paris
  - Hôpital Robert debré, Paris
  - CHU de Rouen, Rouen

REFERENCES:
- [Derived] Lachassinne E, de Pontual L, Caseris M, Lorrot M, Guilluy C, Naud A, Dommergues MA, Pinquier D, Wannepain E, Hausherr E, Jung C, Gajdos V, Cohen R, Zahar JR, Brichler S, Basmaci R, Boelle PY, Bloch-Queyrat C, Aupiais C; COVIDOCRECHE collaborators. SARS-CoV-2 transmission among children and staff in daycare centres during a nationwide lockdown in France: a cross-sectional, multicentre, seroprevalence study. Lancet Child Adolesc Health. 2021 Apr;5(4):256-264. doi: 10.1016/S2352-4642(21)00024-9. Epub 2021 Feb 8. PMID 33571450